CLINICAL TRIAL: NCT06487247
Title: Supportive Transfusion Program for Patients With Hematologic Malignancies: A Cluster Randomized Trial
Brief Title: HEME Home Transfusion Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Oreofe Odejide, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-040; 1R37CA289639 (NIH)
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Myeloma; Myelodysplastic Syndromes; Hematologic Malignancy; Hematologic Diseases; Lymphoma
Keywords: Leukemia; Myeloma; Myelodysplastic Syndromes; Hematologic Malignancy; Hematologic Diseases; Lymphoma
MeSH Terms: conditions — Leukemia; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hematologic Neoplasms; Hematologic Diseases; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Access to home blood transfusions while enrolled in hospice (HEME-Hospice care) (Experimental): Participants assigned to access to HEME-Hospice care who enroll in hospice will have at least once weekly assessment of symptoms of anemia and thrombocytopenia by the study team and will receive transfusions at home as indicated. Individualized care appointments with hospice care team providers, and frequency of visits are determined by individual participant need.
  Interventions: Behavioral: HEME-Hospice Program
- Arm 2: Usual Care (No Intervention): Participants assigned to usual care will receive standard oncology care delivered by the hematologic oncologists. Participants will have access to regular/standard hospice care if they elect to enroll in hospice.

INTERVENTIONS:
Behavioral: HEME-Hospice Program — A care delivery program that combines home-based transfusions with routine home hospice care. Transfusions are administered by trained transfusion nurses. Standard hospice care is provided by an interdisciplinary team of non-transfusion nurse case managers, hospice aides, social workers, and chaplains.
  Other Names: HEME-Hospice
  Arms: Arm 1: Access to home blood transfusions while enrolled in hospice (HEME-Hospice care)

SUMMARY:
This research study is evaluating whether a new care delivery program that provides access to home blood transfusions in hospice (i.e, HEME-Hospice) compared to regular standard of care improves quality of life, mood, and end-of-life health care utilization for patients with hematologic malignancies.

DETAILED DESCRIPTION:
Lack of access to blood transfusions is a key barrier to timely hospice use for patients with blood cancers. Refractory anemia and thrombocytopenia are common for patients with blood cancers and result in debilitating fatigue, shortness of breath, and bleeding. Transfusions palliate these symptoms and improve quality of life (QOL); yet, most hospices do not provide access to transfusions. Patients are thus faced with the agonizing choice of preserving access to vital palliative transfusions versus accessing quality home-based hospice care. Patients with blood cancers and their caregivers report that transfusions are vital for their quality of life, and that access to transfusions is a key factor in deciding whether to opt for hospice care.

The study team has thus developed a new model of care (HEME-Hospice) that provides access to palliative home transfusions to patients with hematologic malignancies who are enrolled in hospice. The purpose of this study is to determine whether access to HEME-hospice versus usual care improves hospice enrollment rates, quality of life (QOL), mood, and end-of-life healthcare utilization for patients with hematologic malignancies as well as QOL and mood of their caregivers. This study is a cluster randomized trial in which hematologic oncologists will be randomly assigned to access to HEME-Hospice versus usual care. Participants in this study will have access to HEME-hospice or usual care based upon the strategy to which their hematologic oncologist has been assigned.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

* Diagnosis of a relapsed/refractory hematologic malignancy
* Age ≥ 18 years
* Receipt of primary oncologic care at DFCI (at least 2 outpatient visits in 12 months prior to enrollment)
* Has received at least one red blood cell (RBC) or platelet transfusion since blood cancer diagnosis in the clinic or hospital setting without a severe transfusion reaction
* Patient resides within catchment served by Care Dimensions Hospice
* Physician-estimated prognosis of six months or less

Inclusion Criteria for Caregivers:

* Identified informal caregiver of enrolled patient with hematologic malignancy
* Age ≥ 18 years

Exclusion Criteria for Patient Participants:

* Age < 18 years
* Already enrolled in hospice
* Resides in nursing home or assisted living facility
* History of previous serious adverse transfusion reaction

Exclusion Criteria for Caregivers:

-Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Hospice Enrollment Rate | 6 months
  Establish that hospice enrollment rate is higher with access to HEME-Hospice versus usual care.
Length of Hospice Enrollment | 6 months
  Number of days from hospice enrollment to date of death or hospice disenrollment

SECONDARY OUTCOMES:
Chemotherapy Utilization in the Last 14 Days of Life | Last 14 days of life
  Compare chemotherapy use in the last 14 days of life between those with access to HEME-Hospice versus usual care
Hospitalization Rate | Last 30 days of life
  Compare hospitalization (2 or more hospitalizations) in the last 30 days of life between those with access to HEME-Hospice versus usual care
Intensive care unit (ICU) Admission Rate | Last 30 days of life
  Compare ICU admission in the last 30 days of life between those with access to HEME-Hospice versus usual care
Hospital Death | Last 30 days of life
  Compare occurrence of death in the hospital between those with access to HEME-Hospice versus usual care
High-Intensity Healthcare Utilization expenditures in the Last 30 Days of life | Last 30 days of life
  Compare the dollar amount of total expenditures between participants with access to HEME-Hospice versus usual care in the final 30 days of life.
Patient Quality of life | 6 months
  Assess whether access to HEME-Hospice is superior to usual care with respect to patient-reported quality of life (QOL) as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Pal version 4.
  Higher scores on the FACIT-Pal version 4 (range 0-184) indicate better QOL.
Functional Assessment of Cancer Therapy-Anemia (FACT-An) Score | 6 months
  Assessed by the FACT-Anemia version 4 subscale, a 20-item survey rated on a 5-point Likert-type scale. Score range is from 0 to 80 with higher scores indicating better quality of life with respect to symptoms related to anemia and fatigue.
Functional Assessment of Cancer Therapy-Thrombocytopenia (FACT-Th6) Score | 6 months
  Assessed by the FACT-Thrombocytopenia version 4 subscale, a 6-item survey rated on a 5-point Likert-type scale. Score range is from 0 to 24 with higher scores indicating better quality of life with respect to thrombocytopenia-related symptoms.
Patient Anxiety Symptoms | 6 months
  Compare anxiety symptoms between patients with access to HEME-Hospice versus usual care, using the Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS) questionnaire.
  Higher scores on the HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Patient Depression Symptoms | 6 months
  Compare depression symptoms between patients with access to HEME-Hospice versus usual care, using the Depression Subscale of the Hospital Anxiety and Depression Scale (HADS) questionnaire.
  Higher scores on the HADS depression subscale (range 0-21) indicate greater depression symptoms.
Caregiver Quality of Life | 6 months
  Assess whether access to HEME-Hospice is superior to usual care with respect to caregiver-reported quality of life (QOL) as measured by the Caregiver Oncology QOL questionnaire.
  Higher scores on Caregiver Oncology QOL instrument (range 0-100) indicate better QOL.
Caregiver Anxiety Symptoms | 6 months
  Compare anxiety symptoms between caregivers with access to HEME-Hospice versus usual care, using the Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS) questionnaire.
  Higher scores on the HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Caregiver Depression Symptoms | 6 months
  Compare depression symptoms between caregivers with access to HEME-Hospice versus usual care, using the depression Subscale of the Hospital Anxiety and Depression Scale (HADS) questionnaire.
  Higher scores on the HADS depression subscale (range 0-21) indicate greater depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Oreofe Odejide, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu